CLINICAL TRIAL: NCT01380652
Title: Effects of Whole Body Vibration Training on Physical Activity in Chronic Obstructive Pulmonary Disease (COPD) III/IV-Patients During a Three-week Rehabilitation
Brief Title: Vibration Training in Chronic Obstructive Pulmonary Disease (COPD)-Patients During a Three-week Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, MD, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGL-Ga-SW-0810
Record Dates: First submitted 2011-04-01; First posted 2011-06-27 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD III/IV; Activity Monitoring; SenseWear; Vibration training; Galileo; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rehabilitation with vibration training (Experimental)
  Interventions: Procedure: whole body vibration training
- rehabilitation without vibration training (No Intervention)

INTERVENTIONS:
Procedure: whole body vibration training — pulmonary rehabilitation with strength and endurance training and additionally vibration training
  Other Names: whole body vibration; Galileo
  Arms: rehabilitation with vibration training

SUMMARY:
The aim of this study is to investigate the change of physical activity in COPD-patients performing a whole body vibration training additional to a standard three-week rehabilitation program in comparison to patients performing merely a standard rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Chronic obstructive pulmonary disease III/IV

Exclusion Criteria:

* Severe exacerbations in the last 4 weeks prior to begin of study (definition of exacerbation: symptoms on more than 3 days with a relevant change in drug therapy (cortisone, antibiotics))
* Severe disease other than COPD, that could influence the results of the study
* Abuse of alcohol or drugs
* Simultaneously participation in another study
* Tachypnea (>30/min)
* Severe exacerbation during rehabilitation
* Cardiac insufficiency (NYHA IV)
* Myocardial infarction during the last 6 weeks
* Mental-health problem
* Pregnancy
* Known HIV-infection
* Slipped disk
* Acute discopathy
* Acute thrombosis
* Implants in trained regions of the body (lower extremities)
* Acute inflammation of the locomotor system, active arthrosis or rheumatoid arthritis
* Acute tendinopathy in trained regions of the body
* Acute hernia
* Fresh fractures, wounds or scars in trained regions of the body
* Gallstones or stones in the urinary tract collection system

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Activity | day 2 and 17
  change in activity from baseline to day 17

SECONDARY OUTCOMES:
Diffusion Capacity | day 1
BODE-Score | day 1 and 19
  Changes in Bode-Score from baseline to day 19
lung function | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Berchtesgadener Land, Schön Kliniken, Schönau am Königssee, Germany